CLINICAL TRIAL: NCT01413048
Title: Phase III Clinical Trial to Evaluate the Antihypertensive Effect of AGSCT101 Versus Carvedilol in Patient With Stage 1 to 2 Essential Hypertension
Brief Title: Clinical Trial to Evaluate the Antihypertensive Effect of AGSCT101 in Patient With Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Woohyuk Jeong/Senior Researcher, Project Planning and Development Team
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1001AGCVSP3
Record Dates: First submitted 2011-08-07; First posted 2011-08-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Essential Hypertension
Keywords: Essential Hypertension; Hypertension
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AGSCT101 (Experimental)
  Interventions: Drug: AGSCT101 12.5mg
- Carvedilol (Active Comparator)
  Interventions: Drug: Carvedilol 25mg

INTERVENTIONS:
Drug: Carvedilol 25mg — Tablet, q.d.
  Arms: Carvedilol
Drug: AGSCT101 12.5mg — Tablet, q.d.
  Arms: AGSCT101

SUMMARY:
The purpose of this study is to evaluate the antihypertensive effect of AGSCT101 tablet in patient with stage 1 to 2 essential hypertension.

DETAILED DESCRIPTION:
This study is 2,8 weeks, multi-center, randomized, double-blind, active clinical trial to evaluate the efficacy and safety of AGSCT101 versus Carvedilol in patient with stage 1 to 2 essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients ≥ 19 years of age
* Mild to moderate essential hypertension: sDBP 90 ~ 109, sSBP 140 ~ 179
* Subjects who agree to participate in this sudy and give written informed consent
* Subjects considered to understand the study, be cooperative, and able to be followed-up until the end of the study

Exclusion Criteria:

* The sitting DBP is more than 110mmHg or the sitting SBP over 180mmHg
* Patients with postural hypotension
* Patients with severe renal(Creatinine more 1.5mg/dl), gastrointestinal, hematological or hepatic(AST, ALT more 3 times more than upper limit of normal)disease
* Female of childbearing potential who does not undergo hysterectomy or is not post-menopausal
* Patients judged to have a history of alcohol or drug abuse by the investigator
* Patients with a history of myocardial infarction, severe coronary artery disease or clinically significant heart failure or valvular defect in last 6 months
* Patients with uncontrolled diabetes mellitus
* Patients participated other clinical trial 12 weeks before Screening Patients judged to be inappropriate for this study by the investigator with other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-03 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure (DBP) | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in diastolic blood pressure (DBP) | 2 weeks
Change from baseline in systolic blood pressure (SBP) | 2, 8 weeks
Proportion of patients who reach overall blood pressure control (defined as BP <140/90) | 8 weeks
Incidence of adverse effects | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Bae Seung, Professor, Principal Investigator — The Catholic University of Korea-St. Mary's Hospital; Hun-Sik Park, Professor, Principal Investigator — Kyungpook National University Hospital; Chang-Gyu Park, Professor, Principal Investigator — Korea University Guro Hospital; Moo-Yong Rhee, Professor, Principal Investigator — Dongguk University Medical Center; Dong-Ju Choi, Professor, Principal Investigator — Seoul National University Bundang Hospital; Seung-Jea Tahk, Professor, Principal Investigator — Ajou University School of Medicine; Jung-Han Yoon, Professor, Principal Investigator — Wonju Christian Hospital; Sung-Ha Park, Professor, Principal Investigator — Severance Hospital; Myung-Ho Jeong, Professor, Principal Investigator — Chonnam National University Hospital; Sang-Wook Kim, Professor, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- The Catholic University of Korea-St. Mary's Hospital, Seoul, South Korea